CLINICAL TRIAL: NCT06958224
Title: Theranostic Approach by Early Multigene Sequencing in Advanced Poor Prognosis Cancers, Not Eligible for Initial Sequencing in Clinical Routine and Selected From the First Line in Molecular Tumour Board.
Brief Title: Theranostic Approach by Early Multigene Sequencing in Advanced Poor Prognosis Cancers
Acronym: ESCAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2023_0285
Record Dates: First submitted 2025-04-16; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Liver Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: Poor prognosis cancers; Multi-gene sequencing; Molecular Tumour Board; Personalized medicine; Clinical trials
MeSH Terms: conditions — Breast Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large and early multigene sequencing (Experimental)
  Interventions: Genetic: Large and early multigene sequencing
- Large Sequential multigene sequencing according to Plan France Medecine Genomique 2025 (Active Comparator)
  Interventions: Genetic: Large and early multigene sequencing

INTERVENTIONS:
Genetic: Large and early multigene sequencing — Part 1 sequential multi-gene sequencing (Simple NGS),
  * Multi-gene DNA sequencing (43 genes panel corresponding to the most frequently targeted molecular alterations)
  * And if no contributive:
  Part 2: randomized study between two sequential approaches
  - Experimental arm: early Multi-gene DNA sequencing (638 genes panel) Multi-gene RNA sequencing (ARCHER panel)
  1. MMR status in molecular biology
  2. - Tumour Mutational Burden
     * Control arm: after 1st line escape, according to Plan France Medecine Genomique 2025 In the Part 2, a new biopsy could be proposed if necessary

SUMMARY:
The European Society for Medical Oncology (ESMO) strongly recommends to develop multigene sequencing in the framework of molecular screening programmes, in order to improve access to innovative drugs and to accelerate clinical research in cancers.

* Accordingly, this project aims to study the contribution of early systematic multigene sequencing (NGS) discussed in Molecular Tumour Board for poor prognosis cancers, with no current indication for early sequencing.
* The investigators teams propose to perform a randomized study in tumours in which actionable therapeutic targets according to the ESMO ESCAT scale are known (ESCAT II/IV) especially in pancreatic ductal adenocarcinoma, hepatocellular carcinoma or triple negative breast cancer.

Two approaches will be compared: a large multigenic early sequencing approach since the first line setting versus a Plan France Medecine Genomique 2025 approach since the second line setting.

The frequency of really initiated therapeutic proposals according to the molecular status will be compared in each group.

DETAILED DESCRIPTION:
Part 1 sequential multi-gene sequencing (Simple NGS),

* Multi-gene DNA sequencing (43 genes panel corresponding to the most frequently targeted molecular alterations)
* And if no contributive:

Part 2: randomized study between two sequential approaches

- Experimental arm: early Multi-gene DNA sequencing (638 genes panel) Multi-gene RNA sequencing (ARCHER panel)

1. MMR status in molecular biology
2. - Tumour Mutational Burden

   * Control arm: after 1st line escape, according to Plan France Medecine Genomique 2025 In the Part 2, a new biopsy could be proposed if necessary

ELIGIBILITY:
Inclusion Criteria:

* - Age >18 years.
* Advanced disease status ("unresectable" or "metastatic").
* Patient included either at the time of diagnostic investigation or during first line of treatment.
* Good general conditions, still compatible with a therapeutic proposal, WHO 0-1.
* The following tumour sites, with poor prognosis and for which ESCAT II/IV treatment targets can be found according to ESMO:

  * pancreatic adenocarcinoma
  * hepatocellular carcinomas,
  * triple negative breast cancer.
* Tumour tissue a priori available in sufficient quantity: at least one biopsy from a visceral metastatic site or surgical specimen (if available) for eligible cancers.
* Patient covered by a social sercurity scheme

Exclusion Criteria:

* - General condition WHO >1 and/or nutritional status not compatible with a therapeutic proposal
* Limiting systemic cardiovascular, renal, bronchopulmonary or endocrinological comorbidities with the initiation of a therapeutic proposal
* Active infection or active chronic disease (diabetes, liver dysfunction, immune disease) making the patient's condition incompatible with a therapeutic proposal.
* A priori unavailable, in insufficient quantity or of suboptimal quality tumour material.
* Administrative reasons: inability to receive informed information, inability to participate in the entire study, lack of social security coverage, refusal to sign consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2028-11-10 (Estimated); Study Completion 2029-01-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of patients receiving a proposal for treatment leading to effective initiation of treatment. | Within 2 years of the first Molecular Tumour Board.

SECONDARY OUTCOMES:
1. Frequency of therapeutic proposals, whether or not leading to treatment, among patients with at least one molecular alteration found | Within 2 years of the first Molecular Tumour Board.
2. The number of potentially targetable molecular alterations found. | Within 2 years of the first Molecular Tumour Board.
The frequency of the types of potentially targetable molecular alterations found according to the ESCAT classification (ESCAT I / II / III / IV). | Within 2 years of the first Molecular Tumour Board.
4. Frequency of types of therapeutic proposals (clinical trials, off-label targeted therapies). | Within 2 years of the first Molecular Tumour Board.
Time to treatment proposal, defined as the time between the date of the first Molecular Tumour Board and the treatment proposal following the second Molecular Tumour Board. | Within 2 years of the first Molecular Tumour Board.